CLINICAL TRIAL: NCT00433264
Title: The Interrelation of the Vasculature, Endothelium, Bone Metabolism and Uremic Toxins in Peritoneal Dialysis
Acronym: INVEST-PD
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Pieter Evenepoel, University Hospitals Leuven
Other Study IDs: ML3645
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Kidney Disease
Keywords: peritoneal dialysis; endothelium; endothelial dysfunction
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Peritoneal Dialysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, DNA
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: peritoneal dialysis — individualised
  Other Names: individualised

SUMMARY:
Despite major advances in the treatment of chronic kidney disease, the age and sex matched mortality far exceeds that of the normal population. As in the normal population, the majority of deaths are related to cardiovascular disease. Mounting data point to the lethal synergy between chronic kidney disease and cardiovascular disease. This relation is present from early stages of chronic kidney disease on.

Several uremic toxins have been demonstrated to play an important role in kidney disease related endothelial dysfunction. In peritoneal dialysis patients, data on the relation between uremic toxins, endothelial dysfunction and microparticles are lacking.

The investigators hypothesize that endothelial dysfunction and uremic toxins are interrelated in peritoneal dialysis patients

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* Maintenance peritoneal dialysis

Exclusion Criteria:

* No informed consent
* Peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary referral center university hospital
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Meijers, MD, Principal Investigator — UZ Leuven; Kathleen Claes, MD, Principal Investigator — UZ Leuven; Pieter Evenepoel, MD, PhD, Study Director — UZ Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium